CLINICAL TRIAL: NCT03581136
Title: Phase II Multi-center Trial Evaluating 5 Fraction S-PBI (Stereotactic Partial Breast Irradiation) for Early Stage Breast Cancer Using the GammaPod
Brief Title: Phase II Multi-center Trial Evaluating 5 Fraction Stereotactic Partial Breast Irradiation Using Gammapod
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Texas Southwestern Medical Center (Other)
Responsible Party: Principal Investigator, Asal Rahimi, MD, University of Texas Southwestern Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: STU 042018-083
Record Dates: First submitted 2018-06-06; First posted 2018-07-10 (Actual); Last update posted 2025-09-29 (Actual); Status verified 2025-09

CONDITIONS: Breast Cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — Chemical Fractionation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (1):
- Prescription Isodose Surface Coverage (Experimental): The dose fractionation to the CTV (1cm expansion on cavity) will be 40Gy/ 5 fractions and the PTV (3 mm expansion of CTV) will be a minimum dose of 30Gy/5 fractions.
  If PTV >100cc or if dose constraints cannot be met on higher dose prescribe CTV (1.0cm) to 35Gy/5 fractions and PTV (3mm) to 30Gy/5 fractions. This is to potentially reduce risk of fat necrosis.
  Interventions: Device: Dose Fractionation

INTERVENTIONS:
Device: Dose Fractionation — Patients will receive 5 fractions of radiation. These should not be on consecutive days. At least 40 hours between each fraction and a maximum of 21 days to complete, i.e.: Tuesday, Thursday, Monday, Wednesday, Friday.

SUMMARY:
Stereotactic radiation has been implemented more than 3 decades ago, initially to radiate benign and later malignant tumors within the brain. Doses up to 24 Gy in one session have been used. Hundreds of thousands of patients have been treated worldwide with very good outcomes . Over the last decade, the stereotactic radiation techniques have been implemented to treat extra-cranial tumors. The challenges of extra cranial tumors were in part target motion during the radiation session, but also accurate re positioning of the patient and of the target volume at time of radiation treatment. Specific immobilization devices are now available to improve accuracy of target localization. Stereotactic radiation therapy is widely available, non-invasive for the patient and less operator dependent as the planning process (from target volume to dose calculation) can be done and verified by different operators through a quality assessment procedure. Stereotactic radiation is a complex type of 3D CRT that is a very attractive technique making the 3D CRT more conformal and more accurate delivery of the prescription dose within the target volume with a very good sparing of surrounding normal tissue. The principles of stereotactic radiation are the following: precise image definition of target volume and OARs, very conformal radiation treatment.

DETAILED DESCRIPTION:
The GammaPod is a new external beam radiotherapy device dedicated for stereotactic radiotherapy of breast cancer (Xcision Medical Systems, LLC, Columbia, Maryland). The design goal of the GammaPod has been the ability to deliver ablative doses with sharp gradients under stereotactic image guidance. Highly focused radiation is achieved at the isocenter due to the cross-firing from 36 radiation arcs generated by rotating 36 individual Cobalt-60 beams.In order to immobilize the breast during imaging and treatment and in order to get a stereotactic localization of the breast target volume, a vacuum-assisted breast immobilization cup with built-in stereotactic frame is used. The patient can be imaged on a CT or MRI wearing the vacuum-assisted breast cup and then be transferred to the GammaPod for treatment. Then, the planner is required to delineate the gross tumor volume (GTV) and its subclinical extensions. Multiple targets within a breast are allowed.Different doses can be prescribed to different targets.One benefit of using the GammaPod over the cyberknife for breast SBRT, is elimination of the need for internal gold fiducial markers, which are required for the cyberknife treatment.

Using a stereotactic technique for APBI allows smaller margins in comparison to a 3DCRT technique. The total expansions on the RAPID trial (3DCRT APBI) were 1.0 cm CTV expansion on the lumpectomy cavity and an additional 1.0 cm for PTV, for a total expansion of 2.0 cm. As a 3DCRT technique was used on the RAPID trial limited number of radiation beams were employed, no Intensity Modulated Radiation Techniques allowed, and the margins used to create a PTV were relatively large (total margin 2 cm).

As the GammaPod will allow us to minimize the volume of normal breast being irradiated, and decrease the PTV volume we hypothesize that a stereotactic technique with the GammaPod will allow us to improve on the 3 year global cosmesis rates (physician and patient) reported in the RAPID trial (3DCRT) by 40% despite 5 daily fractions of SBRT (in contrast to 38.5Gy/10 fractions 3DCRT BID on the RAPID trial) The GammaPod was FDA approved 12-2017.

ELIGIBILITY:
Inclusion Criteria:

Women who satisfy all of the following conditions will be eligible for this study.

1 DCIS or invasive ductal, medullary, papillary, mucinous (colloid), lobular,or tubular histologies.

2. Age ≥ 18 years. 3. ECOG Performance status 0-2. 4. Women of child-bearing potential must agree to use adequate contraception (barrier method of birth control- condom or diaphragm and spermicidal foam; intrauterine device, prescription birth control pills, or abstinence) prior to study entry, for the duration of study participation, and for 90 days following completion of therapy. Should a woman become pregnant or suspect she is pregnant while participating in this study, she should inform her treating physician immediately.

4.1. A female of child-bearing potential is any woman (regardless of sexual orientation, having undergone a tubal ligation, or remaining celibate by choice) who meets the following criteria:

* Has not undergone a hysterectomy or bilateral oophorectomy; or
* Has not been naturally postmenopausal for at least 12 consecutive months (i.e., has had menses at any time in the preceding 12 consecutive months).

  5. Appropriate staging studies identifying as AJCC stage Tis, or T1-T2, N0 (N0i+). The tumor size must be 3 cm or less.

  6. Surgical treatment of the breast with lumpectomy with histologically confirmed margins free of tumor (no ink on margin) for invasive disease, and at least 2mm for Ductal Carcinoma In Situ.. (Re-excision of margins is permitted).

  7. Gross disease within the breast must be unifocal. (Patients with microscopic multifocality are eligible as long as the total extent of tumor, gross and microscopic, occupies a volume with greatest dimension extent of 3 cm or less (regarding the largest diameter of volume occupying space).

  8. Patients with invasive disease are required to have axillary staging including: sentinel node biopsy or axillary dissection. If patients are over age 65, axillary staging is at the discretion of the physician. Patients with DCIS are not required to have axillary staging.

  9. Lymphovascular invasion is allowed if limited or focal.

  10. Ability to understand and the willingness to sign a written informed consent

Exclusion Criteria:

1. Men are not eligible for this study.
2. T2(>3.0 cm), T3, N1, stage III, or stage IV breast cancer
3. Evidence by physical examination or mammography of other suspicious masses, densities, or microcalcifications in either breast, unless biopsied and found to be benign.
4. Patients with non-epithelial breast malignancies such as sarcoma or lymphoma are excluded.
5. Paget's disease of the nipple.
6. Previous thoracic or breast radiation on ipsilateral side. Contralateral breast radiation is not excluded.
7. Treatment plan that includes ipsilateral whole breast or ipsilateral regional nodal irradiation.
8. Any prior treatment with radiation, or chemotherapy (in the neoadjuvant setting) for currently diagnosed breast cancer prior to GammaPod treatment- adjuvant chemotherapy is acceptable.
9. Patients with active collagen vascular disease, specifically dermatomyositis with a CPK level above normal or active skin rash, systemic lupus erythematosis, or scleroderma, or no other exclusions.
10. Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, immunosuppressed patients or psychiatric illness/social situations that would limit compliance with study requirements.
11. Subjects must not be pregnant or nursing due to the potential for congenital abnormalities and the potential of this regimen to harm nursing infants.
12. If the lumpectomy cavity is completely outside of the vacuum assisted breast cup, then patient should not be treated on the GammaPod secondary to concerns of reproducibility.
13. Transplant patients or any patients on immunosuppressive therapy.
14. Breast size that is too large for the breast cup immobilization device.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Men are not eligible for this study.
Enrollment: 74 (Actual)
Dates: Start 2019-04-22 (Actual); Primary Completion 2028-05-25 (Estimated); Study Completion 2030-06-28 (Estimated)

PRIMARY OUTCOMES:
Patient Cosmesis | 3 Years
  To determine the 3 year patient overall global cosmesis score (on scale excellent, good, fair, or poor) and adverse cosmesis using SPBI with the GammPod using a 5 fraction escalated dose regimen (a more hypofractionated regimen compared to conventional APBI regimens). Cosmesis will be determined using patient cosmesis.

SECONDARY OUTCOMES:
Ipsilateral Breast Recurrence Rate | 3 Years
  The definition of treatment failure is histologic evidence of recurrent carcinoma, either invasive or non-invasive (except LCIS) in the ipsilateral breast or chest wall. Clinical evidence of carcinoma by physical examination and/or mammograms will not be construed as evidence of treatment failure without biopsy proof but will be considered as suspicious for recurrence. Ipsilateral breast recurrences will be considered local (infield) if they occur within the prescription isodose volume; they will be considered peripheral if they occur between the prescription isodose volume and a volume 2 cm outside of the prescription isodose volume. Ipsilateral recurrences will be considered non-contiguous or extra field if they are beyond the peripheral volume described above. Exact binomial method will be also used to estimate ipsilateral breast recurrence rate and late toxicity rate along with the corresponding 95% confidence interval.
Disease Specific Survival | 3 Years
  Kaplan-Meier method will be used to estimate disease-specific survival. Specific survival will be measured from the date of study entry to the date of death due to breast cancer. The following will be considered as failure events in assessing disease specific survival:
  Death certified as due to breast cancer.
  Death from other causes with active malignancy.
  Death due to complications of treatment, irrespective of the status of malignancy.
  Death from other causes with previously documented relapse as defined above but inactive at the time of death will not be considered in disease-specific survival, but will be analyzed separately.
Distant Disease-Free Interval | 3 Years
  Defined as the time from registration to first diagnosis of distant disease. The distant disease-free interval will be measured from the date of registration until the date of first diagnosis of distant disease.
Recurrence Free Survival | 3 Years
  Kaplan-Meier method will be used to estimate recurrence-free survival. Time from registration to first diagnosis a local, regional, or distant recurrence.
Treatment Related Toxicity | 18 Months
  To determine treatment related toxicity (Toxicity will be assessed via NCI's Common Toxicity Criteria for Adverse Events (CTCAE) toxicity criteria as well as RTOG-EORTC (Radiation Therapy Oncology Group - European Organization for the Research and Treatment) Late Radiation Toxicity scales.)
Evaluation of Cosmesis from Serial Photography | 3 Years
  Photographs of both breasts will be taken twelve months from the start of therapy and at yearly intervals thereafter up to 3 years after treatment. Digital Photographs will be evaluated using the BCCT.core proprietary software developed by INESC Porto Breast Research Group (50-51) and an independent panel.
Evaluation of Patient Cosmesis | 3 Years
  To determine three year adverse Cosmesis results by an independent expert panel review. Cosmesis will be graded by the patient using the EORTC (European Organization for the Research and Treatment) scale, at baseline, and twelve months from the start of therapy and at yearly intervals thereafter up to 3 years after treatment. Cosmesis forms using the EORTC scale will be completed by the patient.
Physician Cosmesis | 3 Years
  Cosmesis will be graded by the radiation oncologist using the EORTC (European Organization for the Research and Treatment) scale, at baseline, and twelve months from the start of therapy and at yearly intervals thereafter up to 3 years after treatment. Cosmesis forms using the EORTC scale will be completed by physician.

OTHER OUTCOMES:
Health-Related Quality of Life Using EQ-5D | 5 years
  The quality of life questionnaire will be used as a standardized instrument to measure the health outcome. Its provides a simple descriptive profile and a single index value for health status. The US version of the EQ-5D (EuroQol five-dimension scale questionnaire) will be used, to enable mapping of general HR-QOL scores from EQ-5D scores into health state utility scores (ranging from 0 to 100) for the US population. Analyses will be performed for all subjects having received at least one fraction of radiation. The study will use the CTCAE version 5.0 for reporting of acute and late adverse events related to breast will be reported by the physician through exam/assessment during research visit, encompassing events since last research visit. Research will collect and log breast related events for up to 5 years.
Quality of Life Using BREAST-Q | 5 Years
  The BREAST-Q instruments are a series of validated instruments used in the breast cancer population. They will be administered to the patient pre-treatment and at the intervals specified in the Time and Events table. Longitudinal changes in BREAST-Q scores will be characterized, and predictors of adverse scores over time will be evaluated using multivariable analysis. The modules being used are:
  * Satisfaction with breasts
  * Adverse effects of radiation
  * Psychosocial well-being
  * Physical well-being: chest

CONTACTS AND LOCATIONS:
Overall Officials: Asal Rahimi, MD, Principal Investigator — University of Texas Southwestern Medical Center
Locations (2):
- United States (2):
  - University of Maryland Medical Center, Baltimore, Maryland
  - UT Southwestern Medical Centre, Dallas, Texas

IPD SHARING:
Plan to Share IPD: Undecided